CLINICAL TRIAL: NCT04094857
Title: A Phase 1 First-In-Human Study of HBN-1 in Patients Resuscitated Following Out-of-Hospital Cardiac Arrest
Brief Title: Phase 1 Study of HBN-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hibernaid, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBN-1-001-US
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Arrest
Keywords: therapeutic temperature management; therapeutic hypothermia
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Randomized, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HBN-1 Plus Standard of Care (Experimental): Subjects will receive an intravenous loading dose of HBN-1 followed by a 12 hour maintenance infusion plus standard of care targeted temperature management
  Interventions: Drug: HBN-1
- Standard of Care (No Intervention): Subjects will receive standard of care targeted temperature management only

INTERVENTIONS:
Drug: HBN-1 — Intravenous infusion
  Arms: HBN-1 Plus Standard of Care

SUMMARY:
Phase 1 First-in Human randomized, open-label, active control standard of care study of the safety of HBN-1 administered as pharmacologically induced hypothermia as an adjunct to standard of care targeted temperature management in adult patients who have experienced out-of-hospital-cardiac arrest. HBN-1 will be administered IV as a loading dose infusion followed by a 12-hour maintenance infusion.

DETAILED DESCRIPTION:
Phase 1 First-in Human randomized, open-label, active control standard of care study of the safety of HBN-1 administered as pharmacologically induced hypothermia as an adjunct to standard of care targeted temperature management in adult patients who have experienced out-of-hospital-cardiac arrest.

HBN-1 will be administered as an IV solution according to a weight-based escalating loading dose infusion rate scheme involving three sequential cohorts with a loading dose of HBN 1 administered over 60 minutes (Cohort A), 45 minutes (Cohort B), or 30 minutes (Cohort C). For all cohorts, the loading dose will be followed by a 12-hour maintenance infusion of HBN-1.

Dosing cohorts will include a minimum of 6 subjects randomized in a 2:1 ratio of HBN-1 plus standard of care versus standard of care alone. Individual cohorts may be expanded to up to a maximum of 12 subjects . If the cohort is expanded, the additional subjects will receive HBN-1 + SOC.

During the loading dose and maintenance infusion, physical exam, temperature, assessment of shivering, ECG, vital signs, clinical laboratory, blood alcohol level, and neurologic status will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 to 80 years, inclusive
2. Documented diagnosis of OHCA with ventricular tachycardia/fibrillation, asystole or pulseless electrical activity
3. Return of spontaneous circulation within 50 minutes of the event
4. FOUR Motor Score <4
5. Maximum estimated weight not to exceed 100 kg

Exclusion Criteria:

1. Return of spontaneous circulation >8 hours
2. Known history of prior cardiac arrest, alcohol, or substance abuse or dependence
3. Presumed etiology of cardiac arrest is trauma, hemorrhage, or sepsis
4. Comfort measures only or anticipated withdrawal of life-support within 24 hours
5. Is within a protected population group (eg, pregnant or breastfeeding or incarcerated persons)
6. Has history or evidence of significant hepatic dysfunction (Sequential Organ Failure Assessment Hepatic score >2)
7. Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate, e.g. end-stage chronic illness with no reasonable expectation of survival to hospital discharge
8. Is able to obey to verbal commands
9. Is receiving IV vasopressin or lidocaine hydrochloride

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety and recommended Phase 2 loading dose infusion rate of HBN-1 | Initiation of TTM until a minimum of 72 hours
  Safety and tolerability based on evaluation of adverse events, serious adverse events, physical examinations, vital signs measurements, electrocardiograms, and changes in clinical laboratory values (hematology, biochemistry, and urinalysis)

SECONDARY OUTCOMES:
Determine the incidence of the need for implementation of treatment to offset shivering | Initiation of TTM until a minimum of 72 hours
  Number and proportion of subjects who require intervention for shivering.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Katz, MD, Study Director — Hibernaid, Inc; David B Seder, MD, Principal Investigator — MaineHealth
Locations (2):
- United States (2):
  - Maine Medical Center, Portland, Maine
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No